CLINICAL TRIAL: NCT06933615
Title: Development and Evaluation of the Effectiveness of a Mobile Individual Atrial Fibrillation Management (m-BAFY) Program
Brief Title: Mobile Individual Atrial Fibrillation Management Program
Acronym: m-BAFY
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Collaborators: Ege University Hospital (Application and Research Center) (Unknown)
Responsible Party: Principal Investigator, Adile Ay, Lecturer, Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Aay
Record Dates: First submitted 2025-04-02; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Atrial Fibrillation (AF)
Keywords: atrial fibrillation; mobile health; nursing care
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: The universe will consist of all patients diagnosed with AF who apply to the Arrhythmia Polyclinic of the Cardiology Department of Ege University Health Application and Research Center. The sample will consist of patients selected from the universe and who meet the inclusion criteria for the study. Power analysis was performed to determine the number of patients to be included in the study. The power of the test was calculated with the G. Power-3.1.9.2 program. The effect size (d= 0.544) of a similar study in the relevant literature regarding the change in AF-specific quality of life was taken as basis (Woo et al., 2022). Based on this; with an alpha value of 0.05, an effect size of 0.544, and a theoretical power of 0.90, the minimum sample size in the intervention group was calculated as 45 people in total. The groups within the scope of the study were divided into two groups, the intervention group and the control group, using the stratified randomization method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care Group (No Intervention): The standard program of the clinic will be applied to the patients in the control group. No intervention will be made by the researcher. Follow-up data will be collected by the researcher at the first interview and at the end of the 1st and 3rd months using the tools included in the data collection form. At the end of the research, the m-BAFY program will be shared with the patients in the control group.
- The mobile application group (Experimental): Patients in the intervention mobile application group are downloaded to their mobile phones. This application includes information about the patient's disease. Motivational and condition-related messages are sent to their phones.
  Interventions: Other: Training prepared with mobile application

INTERVENTIONS:
Other: Training prepared with mobile application — The m-BAFY program will be loaded onto the mobile phones of patients in the mobile application group. Each patient will be informed on how to use the mobile program. In addition, a short training will be given on how to use the application. With this application, the symptoms and vital signs recorded by the patients will be monitored and individual feedback will be provided. Information on the management of the disease prepared in line with the guidelines is included.
  Arms: The mobile application group

SUMMARY:
The aim of the study is to develop a mobile individual atrial fibrillation management (m-BAFY) program and to evaluate the effects of the program on symptom severity, medication compliance, self-care agency and quality of life. The main questions that the study aims to answer are as follows;

* Is the m-BAFY program effective in symptom control?
* Is the m-BAFY program effective in increasing medication compliance?
* Is the m-BAFY program effective in improving self-care agency?
* Is the m-BAFY program effective in improving quality of life? In order to measure whether m-BAFY is effective, the researchers will download this application to one group's phones, and the other group will not download the application.

Participants;

* Use this application for 3 months
* Patients in the intervention group use the application at least once every two weeks.
* Fill in the symptom diary in the application.
* Clinical interviews are called for the first interview, at the end of the 1st month and at the end of the 3rd month.

DETAILED DESCRIPTION:
The research sample was divided into two groups, the intervention and control groups, using the simple randomization method. The m-BAFY program prepared for the intervention group will be downloaded to their phones and asked to use it for three months. A unique username and password will be created for each patient. Patients' records and navigation between tabs will be tracked via the Firebase system. Motivational messages and feedback will be given to patients. Patients will be informed that they will be provided with consultancy services within the scope of the program content throughout the research.

The standard program of the clinic will be applied to the patients in the control group. No intervention will be made by the researcher. Follow-up data will be collected by the researcher at the end of the 1st and 3rd months using the tools in the data collection form.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years old and above
* Having an AF diagnosis
* Being literate
* Being able to understand and speak Turkish
* Being able to use a smartphone
* Being willing to participate in the study

Exclusion Criteria:

* Hearing and speech problems
* Cardiac surgery < 3 months before the interview date
* Presence of psychiatric disease
* No data entry for at least 2 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-06-10 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
Symptom severity assessed by the University of Toronto Atrial Fibrillation Severity Scale (AFSS) | Baseline, at the end of four weeks and at the end of twelve weeks
  The scale contains three sections, "AF Burden", "Healthcare Use" and "AF Symptom Severity", and a total of 19 items.
Atrial Fibrillation Impact on Quality of Life Questionnaire (AFEQT) | Baseline, at the end of four weeks and at the end of twelve weeks
  The scale consists of 20 items in four sub-dimensions: symptoms, daily activities, treatment anxiety/concern, and treatment satisfaction. A score of zero indicates that the quality of life is negatively affected, while a score of 100 indicates that the quality of life is not negatively affected.
Self-Care Ability Scale | Baseline, at the end of four weeks and at the end of twelve weeks
  The scale consists of 35 items. Each statement is scored from 0 to 4 and answered on a 5-point Likert-type scale. It is ranked as 0 (does not describe me at all), 1 (does not describe me very much), 2 (I have no idea), 3 (describes me a little), 4 (describes me very much). As the score increases, the self-care ability of the patients increases in direct proportion.
Medical Adherence Report Scale | Baseline, at the end of four weeks and at the end of twelve weeks
  It contains five items related to medication compliance. Each item is evaluated on a 5-point Likert type scale where "5=never, 4=rarely, 3=sometimes, 2=often and 1=very often". The lowest score that can be obtained from the scale is 5, and the highest is 25. It is stated that as the score obtained increases, medication compliance increases, and as the score decreases, medication compliance decreases.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No